CLINICAL TRIAL: NCT02509598
Title: A Prospective, Open-Label, Multicenter Study of Lymphoseek® as a Lymphoid Tissue Targeting Agent in Pediatric Patients With Melanoma, Rhabdomyosarcoma, or Other Solid Tumors Who Are Undergoing Lymph Node Mapping
Brief Title: A Study of Lymphoseek® as a Lymphoid Tissue Targeting Agent in Pediatric Patients With Melanoma, Rhabdomyosarcoma, or Other Solid Tumors Who Are Undergoing Lymph Node Mapping
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardinal Health 414, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-18
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Rhabdomyosarcoma; Melanoma
MeSH Terms: conditions — Rhabdomyosarcoma; Melanoma | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran; iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tc99m tilmanocept and Vital Blue Dye (optional) (Experimental): 0.5 mCi, 50 ug of Tc99m tilmanocept single administration. Optionally, 1-3 mL of vital blue dye, single administration (per institution's standard of care).
  Interventions: Drug: Tc99m tilmanocept; Drug: Vital Blue Dye (optional); Procedure: Lymph Node Mapping

INTERVENTIONS:
Drug: Tc99m tilmanocept — A single dose of 0.5 mCi and 50 ug of Tc99m tilmanocept administered intradermally, peritumorally approximately 15 minutes to 8 hours before surgery
  Other Names: Lymphoseek
Drug: Vital Blue Dye (optional) — A single dose 1-3 mL of vital blue dye (1%) administered intradermally at the start of or during surgery (optional, per institution's standard of care).
  Other Names: Lymphazurin; Isosulfan Blue
Procedure: Lymph Node Mapping — Intraoperative lymph node mapping will occur 15 minutes to 8 hours after Tc99m tilmanocept injection

SUMMARY:
Open label, non-randomized, multi-center, within-subject comparative study to evaluate the tolerability and the diagnostic utility of Lymphoseek with optional comparison to VBD in pediatric subjects with melanoma, rhabdomyosarcoma, or other solid tumor. Subject age will range from neonatal through 17 years.

ELIGIBILITY:
Inclusion Criteria:

* The subject's parent(s)/legal guardian(s) understand(s) and voluntarily signed an informed consent document prior to any study-related assessments/procedures being conducted. Where locally applicable, the subject also understands and voluntarily provides his/her assent prior to any study-related assessments/procedures being conducted
* Subject has been diagnosed with melanoma, rhabdomyosarcoma, or other tumor where tumor resection or biopsy is planned and lymph node mapping is appropriate
* The subject is clinically node negative (cN0) at the time of screening
* Age < 18 years
* Male subjects of childbearing potential must be willing to use a condom during sexual intercourse and shall not father a child during the course of the study or will practice complete abstinence while on study
* Female subjects of childbearing potential must agree to the use of two physician-approved contraceptive methods simultaneously or practice complete abstinence while on study

Exclusion Criteria:

* The subject has had preoperative radiation therapy
* Has had previous surgery or radiation to node basins that would be involved in the intraoperative lymph node mapping (ILM) procedure
* Has a known allergy to dextran or VBD (if intended to be used)
* Has a history of alcohol abuse or alcohol dependency in the 3 years before study entry, or is an alcoholic or drug addict, as determined by the investigator
* Before the administration of Lymphoseek, has received any radiopharmaceutical within 7 radioactive half-lives of that radiopharmaceutical

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Cardinal Health 414, LLC
Locations (6):
- United States (6):
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Nemours Children's Hopsital, Orlando, Florida
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Tumor type [Count of Participants; unit: Participants]
  Melanoma | 5
  Rhabdomyosarcoma | 4
  Other solid tumors | 14

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Lymph Nodes Identified Intraoperatively Per Subject
Time Frame: 1 Day
Measure: Mean (95% Confidence Interval); unit: nodes per subject
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
nodes per subject | 3.30 [1.95 to 4.65]

2. Primary Outcome: Subject Localization Rates
Description: The proportion of subjects with Lymphoseek-identified lymph nodes
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
Participants | 22

3. Secondary Outcome: Proportion of Subjects Who Underwent Preoperative SPECT or SPECT/CT
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
Participants | 21

4. Secondary Outcome: Proportion of Subjects With a Lymph Node Identified Preoperatively Using SPECT or SPECT/CT
Time Frame: 1 day
Population: Number of subjects who underwent preoperative SPECT/CT
Measure: Count of Participants; unit: Participants
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 21
Participants | 20

5. Secondary Outcome: Average Number of Lymph Nodes Identified Preoperatively Using SPECT or SPECT/CT Per Subject
Time Frame: 1 Day
Measure: Mean (95% Confidence Interval); unit: nodes per subject
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 21
nodes per subject | 2.75 [1.81 to 3.68]

6. Secondary Outcome: Agreement of the Number of Nodes Identified by Preoperative SPECT or SPECT/CT to Intraoperative Localization
Description: Average difference in number of LNs identified preoperatively with SPECT/CR and number of LNs identified intraoperatively per subject
Time Frame: 1 Day
Measure: Mean (95% Confidence Interval); unit: nodes per subject
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 21
nodes per subject | -0.86 [-2.60 to 0.89]

7. Secondary Outcome: Upstaging
Description: The proportion of patients with pathology-positive lymph nodes who had at least one pathology-positive lymph node that was identified by Lymphoseek and had no other pathology-positive lymph nodes (i.e., identified by any other method)
Time Frame: 1 Day
Population: Number of subjects with pathology-positive nodes
Measure: Count of Participants; unit: Participants
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 2
Participants | 2

8. Secondary Outcome: Nodal False Negative Rate for Nodes Identified
Description: The number of pathology-positive lymph nodes that were missed intraoperatively by mapping agent divided by the total number of pathology-positive lymph nodes for that mapping agent. Population is all subjects with pathology-positive nodes. False negative rate represents the failure rate of the mapping agent to identify sentinel lymph nodes.
Time Frame: 1 Day
Population: Subjects with pathology-positive nodes
Measure: Number (95% Confidence Interval); unit: proportion
Units Other Than Participants: pathology-positive nodes
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 2
Number analyzed (pathology-positive nodes) | 4
proportion | 0 [0 to 0.60]

9. Secondary Outcome: Nodal Sensitivity
Description: The number of pathology-positive lymph nodes that were identified intraoperatively by mapping agent divided by the total number of pathology-positive lymph nodes for that mapping agent. Population is all subjects with pathology-positive nodes. Sensitivity rate represents the success rate of the mapping agent to identify sentinel lymph nodes.
Time Frame: 1 Day
Population: Subjects with pathology-positive nodes
Measure: Number (95% Confidence Interval); unit: proportion
Units Other Than Participants: pathology-positive nodes
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 2
Number analyzed (pathology-positive nodes) | 4
proportion | 1.00 [0.39 to 1.00]

10. Secondary Outcome: Nodal Agreement of Central Pathology Assessment With Local Pathology Assessment of the Excised Lymph Node(s) to Confirm the Presence/Absence of Tumor Metastases
Description: Number of nodes whose local and central pathology results agree divided by the number of nodes with nonmissing local and central pathology results
Time Frame: 1 Day
Measure: Count of Units; unit: Nodes with nonmissing pathology
Units Other Than Participants: Nodes with nonmissing pathology
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
Number analyzed (Nodes with nonmissing pathology) | 58
Nodes with nonmissing pathology | 57

11. Secondary Outcome: Change in Subject Nodal Staging Before and After Surgery Based Upon Nodes Identified
Description: Change in subject nodal staging was assessed via shift tables to show the number of subjects with each combination of presurgery and postsurgery nodal staging. Presurgery staging was based on standard-of-care clinical assessment. Postsurgery staging was based on the pathology results of the nodes identified.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
Participants | 3

12. Secondary Outcome: Number of Changes in Postsurgical Treatment Plan in Relation to Nodes Identified by Lymphoseek
Description: Changes to postsurgical treatment plan will be compared to baseline treatment plan.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
Number analyzed (Participants) | 23
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events beginning on the day of injection through the follow-up assessment (4- to 14-day or 62 ± 7 day, depending on protocol amendment at time of enrollment) were to be reported.
Description: Adverse events, blood samples, physical exam, vital signs and ECGs were collected and monitored at protocol-specified times.
Arm/Group | Tc99m Tilmanocept and Vital Blue Dye (Optional)
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tc99m Tilmanocept and Vital Blue Dye (Optional) (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 2 (4)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1)
pyrexia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tc99m Tilmanocept and Vital Blue Dye (Optional) (N=23)
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT02509598/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT02509598/ICF_001.pdf